CLINICAL TRIAL: NCT05302908
Title: Identifying and Addressing Critical Social, Ethical, and Behavioral Factors Associated With COVID-19 Testing and Vaccination Among Spanish Speakers
Brief Title: COVID-19 Testing and Vaccination Among Spanish Speakers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00079510; 5U01MD017431 (NIH)
Record Dates: First submitted 2022-03-29; First posted 2022-03-31 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: COVID-19; Vaccinations
Keywords: COVID-19; Vaccinations; Spanish-speaking; Latinx; Hispanic/Latino populations
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NuestraSaludSegura intervention (Experimental): Intervention-group Navegantes will be trained and supported for 6 months of implementation in Years 1-2
  Interventions: Behavioral: NuestraSaludSegura
- delayed NuestraSaludSegura intervention (Experimental): delayed-intervention group Navegantes will be trained in Year 2
  Interventions: Behavioral: NuestraSaludSegura

INTERVENTIONS:
Behavioral: NuestraSaludSegura — It blends peer navigation and mHealth

SUMMARY:
Latinx communities are disproportionately affected by the COVID-19 pandemic, with Spanish-speaking Latinx communities carrying even heavier burdens of infection, hospitalization, and mortality. Major barriers to COVID-19 testing and vaccination exist, and a profound need remains to understand and address the social, ethical, and behavioral implications (SEBI) of COVID-19 testing and vaccination within Latinx communities. Our community-academic partnership proposes a rigorous mixed-methods, community-based participatory research study to better understand the SEBI of COVID-19 testing and vaccination and to refine and test a novel and culturally congruent intervention that integrates two evidenced-based strategies - peer navigation and mHealth - to increase COVID-19 testing and vaccination within Spanish-speaking Latinx communities.

DETAILED DESCRIPTION:
A profound need remains to understand the social, ethical, and behavioral implications (SEBI) of COVID-19 testing and vaccination interventions within Spanish-speaking Latinx communities. The proposal is a conceptually integrated community-based participatory research (CBPR) study that includes systematic data collection on the multilevel factors that influence COVID-19 testing and vaccination; refinement of an efficacious intervention that uses complementary theory-based strategies (i.e., peer navigation and mHealth); intervention implementation and evaluation using a longitudinal group-randomized trial design; and dissemination of findings.

ELIGIBILITY:
Inclusion Criteria: To be eligible to participate in the in the NuestraSaludSegura intervention as a Navegante:

* participant must self-identify as Hispanic/Latinx
* participant must be Spanish speaking
* participant reports having been vaccinated against COVID-19
* participant must be ≥18 years of age
* participant must provide informed consent

Inclusion Criteria: To be eligible to participate in the interviews as a Social Network Member:

* participant must self-identify as Hispanic/Latinx
* participant must be Spanish speaking
* participant must be ≥ 18 years of age
* participant must provide informed consent

Exclusion Criteria:

* less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Rhodes, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rhodes SD, Tanner AE, Mann-Jackson L, Alonzo J, Hall MA, Bertoni AG, McCoy TP, Aguilar-Palma SK, Garcia M, Miranda D, Turner MJ. Increasing COVID-19 testing and vaccination among Spanish speakers in the USA: protocol for the development and evaluation of the Nuestra Comunidad Saludable intervention using a group-randomised trial design. BMJ Open. 2022 Nov 16;12(11):e066585. doi: 10.1136/bmjopen-2022-066585. PMID 36385019

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 274 that enrolled, 266 completed baseline data collection. This is because our Aim 1 Qualitative focused phase of interviews and focus group participants did not all fill out REDCap-based surveys with structured demographic questions. Specifically, 62 of 64 (97%) focus group participants and 24 of 30 (80%) interview participants provided demographic data and are reported below.
Groups:
- Aim 1: Interviews: In-depth interviews with 30 representatives from health and service organizations.
- Aim 1: Focus Group Only: 7 focus groups with 64 diverse adult Spanish-speaking Latine persons.
- Aim 2: NuestraSaludSegura Intervention: Aim 2: NuestraSaludSegura Intervention. This group participated in the study developed Nuestra Salud Segura intervention arm.
- Aim 2: Delayed NuestraSaludSegura Intervention: Aim 2: Delayed NuestraSaludSegura Intervention. Participants in this arm comprised a comparison group until intervention was over, at which the intervention was given (i.e., delayed intervention arm).
Period: Overall Study
Arm/Group | Aim 1: Interviews | Aim 1: Focus Group Only | Aim 2: NuestraSaludSegura Intervention | Aim 2: Delayed NuestraSaludSegura Intervention
Started | 30 (In-depth interviews with 30 representatives from health and service organizations.) | 64 (7 focus groups with 64 diverse adult Spanish-speaking Latine persons.) | 90 | 90
Completed | 30 | 64 | 88 | 89
Not Completed | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Aim 1: Focus Group Only: Aim 1: Focus group only. In-depth interviews with 30 representatives from health and service organizations and 7 focus groups with 64 diverse adult Spanish-speaking Latine persons. Demographic data was provided from 62 of 64 (97%) focus group participants and 24 of 30 (80%) of interview participants. This group gives the demographic data available from the 62 available focus group participants.
- Aim 1: Interviews: Aim 1: Interviews only. In-depth interviews with 30 representatives from health and service organizations and 7 focus groups with 64 diverse adult Spanish-speaking Latine persons. Demographic data was provided from 62 of 64 (97%) focus group participants and 24 of 30 (80%) of interview participants. This group gives the demographic data available from the 24 available interviews' participants.
- Total: Total of all reporting groups
Arm/Group | Aim 1: Focus Group Only | Aim 1: Interviews | Aim 2: NuestraSaludSegura Intervention | Aim 2: Delayed NuestraSaludSegura Intervention | Total
Number analyzed (Participants) | 62 | 24 | 90 | 90 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: We report baseline survey data from Aim 2 participants in the Intervention and Delayed Intervention arms and separately from. Aim 1 participants that were unique from Aim 2 paritcipants and had baseline survey data.
  years | 40.5 (13.6) | 49.0 (11.6) | 41.0 (14.0) | 42.4 (11.6) | 41.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We report baseline survey data from Aim 2 participants in the Intervention and Delayed Intervention arms and separately from Aim 1 participants that were unique from Aim 2 paritcipants and had baseline survey data. Please note that for sex for the 24 interview participants 1 had missing sex.
  Participants
    number analyzed (Participants) | 62 | 23 | 90 | 90 | 265
    Female | 40 | 19 | 71 | 67 | 197
    Male | 22 | 4 | 19 | 23 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: We report baseline survey data from Aim 2 participants in the Intervention and Delayed Intervention arms and separately from. Aim 1 participants that were unique from Aim 2 paritcipants and had baseline survey data.
  Participants
    Hispanic or Latino | 62 | 19 | 90 | 90 | 261
    Not Hispanic or Latino | 0 | 4 | 0 | 0 | 4
    Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: We report baseline survey data from Aim 2 participants in the Intervention and Delayed Intervention arms and separately from. Aim 1 participants that were unique from Aim 2 paritcipants and had baseline survey data.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 1 | 0 | 2 | 3
    White | 2 | 11 | 16 | 12 | 41
    More than one race | 1 | 1 | 10 | 21 | 33
    Unknown or Not Reported | 59 | 11 | 64 | 55 | 189

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Ever Tested
Description: Number of Subjects Ever Tested
Time Frame: Baseline
Population: Aim 2 had 180 enrolled - 20 Navegantes/Peer Interventionist and 160 participants with 80 per arm. Of the 80 per arm, n=78 completed follow-up for Intervention and n=79 completed follow-up for Delayed Intervention arm.
Measure: Count of Participants; unit: Participants
Arm/Group | NuestraSaludSegura Intervention | Delayed NuestraSaludSegura Intervention
Number analyzed (Participants) | 78 | 79
Participants | 70 | 58

2. Primary Outcome: Number of Subjects Ever Vaccinated
Description: Number of Subjects Ever Vaccinated
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NuestraSaludSegura Intervention | Delayed NuestraSaludSegura Intervention
Number analyzed (Participants) | 78 | 79
Participants | 66 | 64

3. Primary Outcome: Number of Subjects Up to Date on Recommended Doses
Description: Number of Subjects Up to Date on Recommended Doses
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NuestraSaludSegura Intervention | Delayed NuestraSaludSegura Intervention
Number analyzed (Participants) | 78 | 79
Participants | 22 | 13

4. Primary Outcome: Number of Doses Received
Description: Number of Doses Received
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Doses
Arm/Group | NuestraSaludSegura Intervention | Delayed NuestraSaludSegura Intervention
Number analyzed (Participants) | 78 | 79
Number of Doses | 2.6 (1.1) | 2.6 (0.8)

5. Primary Outcome: Number of Subjects Ever Tested
Description: Number of Subjects Ever Tested
Time Frame: Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NuestraSaludSegura Intervention | Delayed NuestraSaludSegura Intervention
Number analyzed (Participants) | 78 | 79
Participants | 70 | 64

6. Primary Outcome: Number of Subjects Ever Vaccinated
Description: Number of Subjects Ever Vaccinated
Time Frame: Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NuestraSaludSegura Intervention | Delayed NuestraSaludSegura Intervention
Number analyzed (Participants) | 78 | 79
Participants | 69 | 67

7. Primary Outcome: Number of Subjects Up to Date on Recommended Doses
Description: Number of Subjects Up to Date on Recommended Doses
Time Frame: Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NuestraSaludSegura Intervention | Delayed NuestraSaludSegura Intervention
Number analyzed (Participants) | 78 | 79
Participants | 37 | 30

8. Primary Outcome: Number of Doses Received
Description: Number of Doses Received
Time Frame: Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Doses
Arm/Group | NuestraSaludSegura Intervention | Delayed NuestraSaludSegura Intervention
Number analyzed (Participants) | 78 | 79
Number of Doses | 3.0 (1.3) | 2.7 (1.0)

ADVERSE EVENTS:
Time Frame: For Aim 1 with both interviews and focus groups, the time frame of collection was from study beginning until study interview/focus group completion, including those who provided REDCap survey data additionally. These data were cross-sectional and not followed/collected over multiple time-points. For Aim 2 RCT with intervention and delayed intervention groups, the time frame of collection was from study beginning (baseline) until immediate post-intervention at 6-months follow-up later.
Arm/Group | Aim 1: Interviews | Aim 1: Focus Group Only | Aim 2: NuestraSaludSegura Intervention | Aim 2: Delayed NuestraSaludSegura Intervention
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/64 | 0/90 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/64 | 0/90 | 0/90
Other Adverse Events (participants affected / at risk) | 0/30 | 0/64 | 0/90 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT05302908/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT05302908/ICF_000.pdf